CLINICAL TRIAL: NCT03643354
Title: Evaluation of the Prevalence of BPPV and Longterm Effects of Its Therapy in Retirement Homes
Brief Title: Evaluation of the Prevalence of BPPV and Longterm Effects of Its Therapy Using the Rotundum Device in Retirement Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: BPPV Retirement Homes
Record Dates: First submitted 2018-08-13; First posted 2018-08-22 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Benign Paroxysmal Positional Vertigo
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of prevalence of BPPV (Experimental): Epley/Barbeque maneuver will be performed using the Rotundum Device to assess if subject has BPPV, patient will thereafter be treated for it using the Rotundum Device.
  Interventions: Diagnostic Test: Epley maneuver/Barbeque maneuver

INTERVENTIONS:
Diagnostic Test: Epley maneuver/Barbeque maneuver — Subjects will be rotated using the Rotundum Device to perform the previously described maneuvers Epley/Barbeque to evaluate the presence of BPPV.

SUMMARY:
Benign paroxysmal positional vertigo (BPPV) is one of the most common types of vertigo, especially in elderly. Therefore the investigators have set the goal to evaluate the prevalence of BPPV and its therapy using the Rotundum device in elderly living in retirement homes. Furthermore the investigators use a questionnaire to evaluate possible predictive signs to improve the diagnosis of this disease.

ELIGIBILITY:
Inclusion Criteria:

* Lives in retirement home/has vertigo/has signed the informed consent

Exclusion Criteria:

* severe heart failure
* untreated cardiac arrythmia
* severe autonomic Dysregulation
* untreated epilepsy
* untreated cervical vertebral body fracture
* inability to follow the test
* weight over 150kg or under 40kg
* height below 140cm or over 200cm
* bedridden
* already participated this study
* participant is connected to the study team

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 2018-11-25 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of BPPV | Subjects (outcome measure) are assessed during the first 4 Years
  subjects

SECONDARY OUTCOMES:
Evaluation of predictive Factors | Is assessed after all subjects have been tested (after 5 Years)
  Questionnaire answers

CONTACTS AND LOCATIONS:
Overall Officials: n6iqtwqp Y Bögli, Principal Investigator — University of Zurich
Locations (1):
- Stefan Yu Boegli, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Muller R, Zangger P, Straumann D, Bogli SY. Dizziness and benign paroxysmal positional vertigo among retirement home residents: a cross-sectional descriptive and interventional study. BMC Geriatr. 2022 Feb 12;22(1):120. doi: 10.1186/s12877-022-02818-w. PMID 35151262